CLINICAL TRIAL: NCT00723437
Title: Evaluation of Nail Psoriasis Severity Index (NAPSI) and Modified Napsi in Patients With Nail Psoriasis Treated With Acitretin
Brief Title: Evaluation of the Efficacy of Acitretin Therapy for Nail Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istituti Fisioterapici Ospitalieri (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Antonella Tosti MD, University of Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NAIL1
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2008-07-28 (Estimated); Status verified 2008-07

CONDITIONS: Psoriasis
Keywords: nail, psoriasis, NAPSI,acitretin
MeSH Terms: conditions — Psoriasis | interventions — Acitretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: acitretin — Acitretin at the dosage of 0.2 to 0.3 mg/Kg/day for 6 months.
  Other Names: Neotigason

SUMMARY:
Objective:

Efficacy of systemic retinoid therapy of nail psoriasis has never been assessed objectively. Evaluate therapeutic efficacy of acitretin in patients with isolated nail psoriasis.

Design:

Open-study on thirty-six patients with moderate to severe nail psoriasis treated with acitretin.

Participants:

Patients included 27 men and 9 women (mean age 41) with nail psoriasis. Intervention: Therapy consisted of acitretin 0.2 to 0.3 mg/Kg/day for 6 months.

Main Outcome Measure(s):

Clinical evaluation, NAPSI and modified NAPSI scores before therapy, every 2 months during therapy and 6 months after treatment.

DETAILED DESCRIPTION:
The Nail Psoriasis Severity Index (NAPSI) has been designed and successfully implemented to grade severity of psoriatic nail disease. Moreover, the utilization of the NAPSI score and a modified version of this severity index score as an instrument to monitor response to therapy has been recently documented in the medical literature .This open study involves thirty-six patients with moderate to severe nail psoriasis treated with low-dose acitretin from January 2005 to January 2007.Acitretin was given at the dosage of 0.2 to 0.3 mg/Kg/day for 6 months. Laboratory investigations and clinical evaluation, which included photographic record and scoring of NAPSI and modified NAPSI, were performed every 2 months. Investigator evaluation was performed using a 0 (no improvement) to 3 (cleared or almost cleared) score Treatment satisfaction by patients and tolerability were assessed at each visit. All patients were followed for at least 6 months after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients with moderate to severe nail psoriasis

Exclusion Criteria:

* premenopausal women
* patients with hepatic, renal or metabolic diseases
* patients with skin or symptomatic arthropathic psoriasis
* previous systemic treatment for nail psoriasis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-01; Primary Completion 2007-01 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
correlate clinical improvement with % reduction in the NAPSI Score | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Tosti, MD, Principal Investigator — University of Bologna
Locations (1):
- Department of Dermatology University of Bologna, Bologna, Italy

REFERENCES:
- [Background] Rich P, Griffiths CE, Reich K, Nestle FO, Scher RK, Li S, Xu S, Hsu MC, Guzzo C. Baseline nail disease in patients with moderate to severe psoriasis and response to treatment with infliximab during 1 year. J Am Acad Dermatol. 2008 Feb;58(2):224-31. doi: 10.1016/j.jaad.2007.07.042. Epub 2007 Dec 20. PMID 18083272
- [Background] Rich P, Scher RK. Nail Psoriasis Severity Index: a useful tool for evaluation of nail psoriasis. J Am Acad Dermatol. 2003 Aug;49(2):206-12. doi: 10.1067/s0190-9622(03)00910-1. PMID 12894066
- [Background] Brazzelli V, Martinoli S, Prestinari F, Borroni G. An impressive therapeutic result of nail psoriasis to acitretin. J Eur Acad Dermatol Venereol. 2004 Mar;18(2):229-30. doi: 10.1111/j.1468-3083.2004.00667.x. No abstract available. PMID 15009317
- [Background] Cassell SE, Bieber JD, Rich P, Tutuncu ZN, Lee SJ, Kalunian KC, Wu CW, Kavanaugh A. The modified Nail Psoriasis Severity Index: validation of an instrument to assess psoriatic nail involvement in patients with psoriatic arthritis. J Rheumatol. 2007 Jan;34(1):123-9. PMID 17216680